CLINICAL TRIAL: NCT03210038
Title: Cystoscopy in Females: Is There a Difference Between Rigid and Flex Cystoscopy, and Does it Require Local Anasthesia?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Prof. Kobi Stav, Senior Urologist, Assaf-Harofeh Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 0290-16-ASF
Record Dates: First submitted 2017-05-21; First posted 2017-07-06 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: Hematuria; Dysuria; Recurrent Uti
Keywords: Cystoscopy
MeSH Terms: conditions — Hematuria; Dysuria; Urinary Tract Infections | interventions — Lidocaine; Water

STUDY DESIGN:
Intervention Model Description: Pain assessment 4 randomly assigned groups of women divided by type of cystoscope and type of local anesthesia.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Rigid cystoscopy, water based gel on introitus (Active Comparator): Rigid cystoscopy, Wolf 17FR. Pad soaked with water based gel put on introitus for 5 minutes prior to procedure.
  Interventions: Drug: Water
- Rigid cystoscopy, esracain gel based on introitus (Active Comparator): Rigid Cystoscopy, Wolf 17FR. Pad soaked with Esracain (Lidocaine) put on the introitus for 5 minutes prior to procedure.
  Interventions: Drug: Lidocaine
- Flexible cystoscopy, water based gel on introitus (Active Comparator): Flexible cystoscopy, Olympus 16FR. Pad soaked with water based gel put on introitus for 5 minutes prior to procedure.
  Interventions: Drug: Water
- Flexible cystoscopy, Esracain gel based on introitus (Active Comparator): Flexible cystoscopy, Olympus 16FR. Pad soaked with Esracain (Lidocaine) put on the introitus for 5 minutes prior to procedure.
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Lidocaine — Pad soaked with lidocaine gel (Esracaine) left on the introitus for 5 minutes
  Arms: Flexible cystoscopy, Esracain gel based on introitus; Rigid cystoscopy, esracain gel based on introitus
Drug: Water — Water based non-anesthetic lubricant gel left on the introitus for 5 minutes.
  Arms: Flexible cystoscopy, water based gel on introitus; Rigid cystoscopy, water based gel on introitus

SUMMARY:
Women arriving to the Urology department outpatient clinic at Assaf-Harofeh Medical Center in order to undergo a cystoscopy examination will be recruited.

Patients will be randomly assigned to one of four groups by method of cystoscopy (flexible and rigid) and by use of anesthesia to the introitus.

Pain levels will be recorded prior to the examination, during entrance of the cystoscope in the urethral meatus, immediately after the examination and 15 minutes after conclusion.

ELIGIBILITY:
Inclusion Criteria:

* All women referred to elective outpatient cystoscopy.

Exclusion Criteria:

* Known urethral stricture.
* Known allergy to lubricant/anesthesia gel.
* Patients under the age of 18 (minors).
* Patients with current Urinary Tract Infections.
* Chronic pelvic pain (e.g Interstitial Cystitis/Bladder Pain Syndrome.
* Known neurlogical or other chronic pain syndrome requiring chronic analgesia medication.
* Mentally incapable for consensual agreement of participation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 120 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Pain before procedure | Before cystoscopy
  Pain measurement using a 0-10 visual analogue scale (VAS) and comparison of average pain score between the four study groups.
Pain during meatus insertion of cystoscope | During the procedure, at the moment of cystoscopy insertion through the urethra
  Pain measurement using a 0-10 visual analogue scale (VAS) and comparison of average pain score between the four study groups.
Pain immediately after procedure | Immediately after withdrawal of the cystoscope from the urethra
  Pain measurement using a 0-10 visual analogue scale (VAS) and comparison of average pain score between the four study groups.
Pain 15 minutes after procedure | 15 minutes after end of procedure
  Pain measurement using a 0-10 visual analogue scale (VAS) and comparison of average pain score between the four study groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Assaf Harofe Medical Center, Be’er Ya‘aqov, Israel

IPD SHARING:
Plan to Share IPD: Yes
IPD data includes age, BMI, previous medical, urological information. Pain levels during different stages of cystoscopy will be recorded.

REFERENCES:
- [Result] Aaronson DS, Walsh TJ, Smith JF, Davies BJ, Hsieh MH, Konety BR. Meta-analysis: does lidocaine gel before flexible cystoscopy provide pain relief? BJU Int. 2009 Aug;104(4):506-9; discussion 509-10. doi: 10.1111/j.1464-410X.2009.08417.x. Epub 2009 Feb 23. PMID 19239453
- [Result] Patel AR, Jones JS, Babineau D. Lidocaine 2% gel versus plain lubricating gel for pain reduction during flexible cystoscopy: a meta-analysis of prospective, randomized, controlled trials. J Urol. 2008 Mar;179(3):986-90. doi: 10.1016/j.juro.2007.10.065. Epub 2008 Jan 18. PMID 18206920
- [Result] Seklehner S, Remzi M, Fajkovic H, Saratlija-Novakovic Z, Skopek M, Resch I, Duvnjak M, Hruby S, Librenjak D, Hubner W, Breinl E, Riedl C, Engelhardt PF. Prospective multi-institutional study analyzing pain perception of flexible and rigid cystoscopy in men. Urology. 2015 Apr;85(4):737-41. doi: 10.1016/j.urology.2015.01.007. PMID 25817101
- [Result] Stav K, Ohlgisser R, Siegel YI, Beberashvili I, Padoa A, Zisman A. Pain during Female Urethral Catheterization: Intraurethral Lubricant Injection versus Catheter Tip Lubrication--A Prospective Randomized Trial. J Urol. 2015 Oct;194(4):1018-21. doi: 10.1016/j.juro.2015.03.097. Epub 2015 Mar 25. PMID 25818032